CLINICAL TRIAL: NCT07281352
Title: Psilocybin-Assisted Cognitive Behavioral Therapy for Depression
Brief Title: RCT of Psilocybin-assisted CBT for Depression
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Marc J. Weintraub, PhD, Assistant Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-2134; R34AT013077 (NIH)
Record Dates: First submitted 2025-12-08; First posted 2025-12-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Diorder
Keywords: psilocybin; cognitive behavioral therapy
MeSH Terms: interventions — Psilocybin; Pharmaceutical Preparations; Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: The study involves randomization of 50 participants (1:1) to either PA-CBT or psilocybin-assisted therapy with minimal therapeutic support.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: Psilocybin + CBT (Experimental): Participants will receive 12 sessions of cognitive-behavioral therapy (CBT) along with two psilocybin-drug sessions -- the first following the third CBT session (10mg of psilocybin, taken orally) and the second following the sixth CBT session (25mg of psilocybin, taken orally).
  Interventions: Drug: Psilocybin (drug); Behavioral: cognitive behavioral therapy
- Psilocybin + Minimal supportive therapy (Active Comparator): Participants will receive 6 sessions of supportive, non-directive therapy along with two psilocybin-drug sessions -- the first following the third therapy session (10mg of psilocybin, taken orally) and the second following the fourth therapy session (25mg of psilocybin, taken orally).
  Interventions: Drug: Psilocybin (drug); Behavioral: Minimal supportive therapy

INTERVENTIONS:
Drug: Psilocybin (drug) — Participants will receive two doses of psilocybin (10mg, 25mg).
Behavioral: cognitive behavioral therapy — Twelve total sessions of therapy, including manualized cognitive behavioral therapy for major depressive disorder, including psychoeducation about depression, cognitive skills, and behavioral skills as well as preparation for psilocybin.
  Arms: Experimental: Psilocybin + CBT
Behavioral: Minimal supportive therapy — Six total therapy sessions. Preparation for psilocybin in the first three sessions plus supportive, nondirective psychotherapy in the final three sessions.
  Arms: Psilocybin + Minimal supportive therapy

SUMMARY:
The primary objectives of this clinical investigation are to (1) determine the acceptability and feasibility of joining psilocybin-assisted therapy with cognitive-behavioral therapy (PA-CBT) for patients with depression, (2) optimize CBT to most effectively integrate the psilocybin experience with psychotherapy and (3) examine the clinical benefit of psilocybin as an adjunct to cognitive-behavioral therapy (CBT) for major depressive disorder.

This study is a randomized, two-arm, fixed dose trial that will test the feasibility, acceptability, and participant and therapist adherence to PA-CBT. Both treatment arms will receive two doses of psilocybin (10mg and then 25mg, separated by one month). In Phase II, participants will be randomized (1:1) to either a 12-session PA-CBT or a 6-session standard psilocybin-assisted therapy (PAT) condition (3 hours of preparation plus 3 hours of supportive therapy integration following the psilocybin experiences).

ELIGIBILITY:
Inclusion Criteria:

* Ages 21-60,

  * Able to swallow capsules,
  * Patients with a current major depressive episode or a history of major depressive episodes based on the DSM-5 criteria (American Psychiatric Association, 2013),
  * Active current depressive symptoms (i.e., scores >16 on the Hamilton-Depression Rating Scale (HAM-D) covering the prior 2 weeks; Hamilton, 1986),
  * Have an identified support person who can pick up the individual from UCLA Semel Institute and drive individual home following psilocybin sessions,
  * For women of child-bearing potential - using one form of highly effective contraception (e.g., oral contraceptive pill) and willingness to continue contraceptive use for duration of study
  * Patient has been medically cleared for the study by a physician.

Exclusion Criteria:

* A personal or family history (first or second-degree) of psychosis or bipolar disorder

  * Resting blood pressure above 140 systolic, 90 diastolic (averaged across four separate measurements)
  * Meeting criteria for a DSM-5 cluster B personality disorder (narcissistic, histrionic, borderline, antisocial personality disorder),
  * Active suicidality (as indicated by a 3 or greater on item 3 of the HAM-D) or other psychiatric disturbance requiring acute treatment
  * Current use of antidepressants or other serotonergic-affecting substances (e.g., St. John's Wort and 5-hydroxytryptophan),
  * Currently receiving cognitive behavioral therapy,
  * Any of the following cardiovascular conditions: uncontrolled hypertension, coronary artery disease, congenital long QT syndrome, cardiac hypertrophy, cardiac ischemia, congestive heart failure, myocardial infarction, tachycardia, artificial heart valve, a clinically significant screening ECG abnormality, or any other significant cardiovascular condition
  * A history of stroke or Transient Ischemic Attack (TIA)
  * Epilepsy or history of seizures
  * Insulin-dependent diabetes
  * Meeting criteria for a DSM-5 substance abuse or dependence within prior 6 months
  * Positive urine drug screen for illicit substances
  * Use of other psychedelics or ketamine within prior 12 months
  * Adverse prior reaction to a psychedelic agent
  * Pregnant, trying to get pregnant, or nursing

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-05 (Actual); Primary Completion 2027-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Client Satisfaction Questionnaire - 8 | 4-month treatment period
  Treatment acceptability as measured by the participant. Total scores range from 8 to 32, with the higher number indicating greater satisfaction.
Retention/Attrition | 4-month treatment period
  Feasibility as measured by the number of participants retained in each treatment condition over the course of the study treatment
Hamilton Depression Rating Scale | 7-month study period
  symptom severity scored from 0-53, with larger values indicating greater depressive severity
Global Assessment of Functioning | 7-month study period
  psychosocial functioning scored from 0-100, with larger values indicating better functioning

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Semel Institute, Los Angeles, California, United States